CLINICAL TRIAL: NCT04745663
Title: Optimizing Preoperative Disinfection of Eyes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not the expected 2/3 but only 1/3 of conjunctiva samples got bacterial growth. Lack of resources to keep the study going with more participants and over a considerably longer time than anticipated.
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SW2019-3; 2019-001179-35 (EudraCT Number)
Record Dates: First submitted 2021-02-05; First posted 2021-02-09 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Eye Infections
Keywords: Disinfection; Pre-operative; Povidone Iodine; Eye surgery
MeSH Terms: conditions — Eye Infections

STUDY DESIGN:
Intervention Model Description: Both eyes of the participants are tested; one eye randomised to receive the intervention and the second eye to receive the standard disinfection.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Povidone-Iodine 0.3 % (Experimental): A tampon is soaked in diluted PI 0.3% and placed on the inside of the lower eyelid of one eye, where it will release iodine molecules for 20 minutes before being removed.
  Interventions: Drug: Povidone-Iodine 0.3%
- Povidone-Iodine 5 % (Active Comparator): Eye drops of 5% PI is the standard disinfection before eye surgery. The drops will be dripped in one eye and allowed to work for 2 minutes.
  Interventions: Drug: Povidone-Iodine 5%

INTERVENTIONS:
Drug: Povidone-Iodine 0.3% — Low concentration iodine
  Arms: Povidone-Iodine 0.3 %
Drug: Povidone-Iodine 5% — Standard concentration iodine
  Arms: Povidone-Iodine 5 %

SUMMARY:
Topical povidone-iodine (PI) is widely used as ocular antiseptic before and after surgery. The standard dose of 5% PI is however, associated with ocular irritation. We therefore want to test if a lower concentration of PI can be similarly efficacious in reducing bacterial growth while reducing ocular irritation.

ELIGIBILITY:
Inclusion Criteria:

* Patients remitted to intravitreal injections at St. Olavs hospital.
* Patients competent to give written consent

Exclusion Criteria:

* Infectious disease
* Known epitheliopathy
* Contact lens wear
* Use of prescription ophthalmic medications
* Diabetes

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Conjunctival bacterial culture | 1 hour. Bacterial sample is taken before and immediately after disinfection
  Change in colony-forming units (CFU) per milliliter (ml)

SECONDARY OUTCOMES:
Patient pain score | During disinfection and after 1 hour when the anesthetic no longer is effective
  Verbal numeric rating scale, from 0 to 10.
Ocular staining score (OSS) | 1 hour after disinfection
  Modified OSS using fluorescein dye

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Helbostad, MD PhD, Study Director — Norwegian University of Science and Technology; Marit Fagerli, MD, Study Director — Clinic of Ear-Nose-Throat, Eye and Maxillofacial Surgery, St. Olavs Hospital
Locations (1):
- St Olavs Hospital, Trondheim, Norway